CLINICAL TRIAL: NCT01972178
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled 12-Week Phase II Proof of Concept Study to Evaluate the Efficacy and Safety of PRC-4016 600 mg Once Daily Versus Placebo in Statin-Stable Subjects With Mixed Dyslipidemia
Brief Title: Efficacy and Safety of PRC-4016 in Subjects With Mixed Dyslipidemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pronova BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTN 4016 13202
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRC-4016 (Experimental): PRC-4016, oral administration once daily, capsule
  Interventions: Drug: PRC-4016; Drug: Statins
- Placebo (Placebo Comparator): Placebo, oral administration once daily, capsule
  Interventions: Drug: Placebo; Drug: Statins

INTERVENTIONS:
Drug: PRC-4016
  Arms: PRC-4016
Drug: Placebo
  Arms: Placebo
Drug: Statins — Any statin allowed (i.e. rosuvastatin, simvastatin, pravastatin, atorvastatin etc)

SUMMARY:
The objective of this study is

* To evaluate the efficacy of PRC-4016 by assessment of the percentage change in blood lipids and lipoprotein parameter from baseline after 12 weeks of treatment
* To evaluate the safety of PRC-4016 as assessed by adverse events and other safety parameters

DETAILED DESCRIPTION:
6-8 weeks screening period with diet/lifestyle stabilization and lipid qualification

ELIGIBILITY:
Main Inclusion Criteria:

* Fasting triglycerides 200-499 mg/dl
* Non-HDL-C > 130 mg/dl
* Stable statin treatment

Exclusion Criteria:

* Type I diabetes or uncontrolled type II diabetes
* Recent cardiovascular or coronary event
* History of pancreatitis
* History or evidence of major and clinically significant diseases that would interfere with the conduct of the study or interpretation of data
* Uncontrolled hypertension

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Percent change in Non-HDL-C from baseline to Week 12 | from baseline to Week 12

SECONDARY OUTCOMES:
Change in triglycerides from baseline to Week 12 | from baseline to Week 12
Change in HDL-C from baseline to Week 12 | from baseline to Week 12
Change in LDL-C from baseline to Week 12 | from baseline to Week 12
Change in VLDL-C from baseline to Week 12 | from baseline to Week 12
Change in total cholesterol from baseline to Week 12 | from baseline to Week 12
Change in ApoA1 from baseline to Week 12 | from baseline to Week 12
Change in ApoB from baseline to Week 12 | from baseline to Week 12
Change in insulin from baseline to Week 12 | from baseline to Week 12
Change in fasting plasma glucose from baseline to Week 12 | from baseline to Week 12
Change in HbA1c from baseline to Week 12 | from baseline to Week 12
Change in Lp-PLA2 from baseline to Week 12 | from baseline to Week 12
Change in hsCRP from baseline to Week 12 | from baseline to Week 12
Change in red blood cell content of EPA and DHA from baseline to Week 12 | from baseline to Week 12
Change in Insulin Resistance (HOMA) from baseline to Week 12 | from baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Pål Nord, MD, MPH, Study Director — Pronova BioPharma
Locations (29):
- United States (29):
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Terence Hart, MD, Muscle Shoals, Alabama
  - Pacific Oaks Medical Group, Beverly Hills, California
  - National Research Institute - Wilshire, Los Angeles, California
  - Research Across America - Santa Ana, Santa Ana, California
  - Encompass Clinical Research, Spring Valley, California
  - Jacksonville Impotence Treatment Center, Jacksonville, Florida
  - Compass Research East, LLC, Oviedo, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Meridien Research, St. Petersburg, Florida
  - Meridien Research- Tampa, Tampa, Florida
  - Evanston Premier Healthcare Research LLC, Evanston, Illinois
  - Medisphere Medical Research Center, Evansville, Indiana
  - Heartland Research Assoc., LLC, Newton, Kansas
  - Louisville Metabolic and Atherosclerosis Research Center (L-MARC), Louisville, Kentucky
  - Troy Internal Medicine, P.C., Troy, Michigan
  - Radiant Research - Edina, Edina, Minnesota
  - Peters Medical Research, High Point, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Sterling Research Group, Ltd. - Auburn, Cincinnati, Ohio
  - Metabolic and Atherosclerosis Research Center, Cincinnati, Ohio
  - Columbus Clinical Research, Inc., Columbus, Ohio
  - PSB Research/P. S. Bains, M.S., D.O., Marion, Ohio
  - RAS Health Ltd, Marion, Ohio
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - Green and Seidner Family Practice Associates, Lansdale, Pennsylvania
  - Padre Coast Clinical Research, Corpus Christi, Texas
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - National Clinical Research - Richmond, Inc., Richmond, Virginia